CLINICAL TRIAL: NCT06713564
Title: A Phase 1b, Single Dose, Open-Label, Dose-escalation Study to Investigate the Safety and Imaging Characteristics of LS301-IT for Intraoperative Imaging of Lung Cancer
Brief Title: A Single Dose, Open-Label, Dose-escalation Study of the Safety and Imaging Characteristics of LS301-IT for Intraoperative Imaging of Lung Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Integro Theranostics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: LS301-IT-B102
Record Dates: First submitted 2024-11-19; First posted 2024-12-03 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Lung Cancers
Keywords: lung cancer imaging; lung cancer surgery
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: A single-dose, open-label, dose-escalation Phase 1b study in patients scheduled to undergo minimally invasive surgery (MIS) for known or suspected lung cancer via thoracoscopy (i.e., VATS). Single dose IV administration of LS301-IT, either on the day before surgery with 4 different doses in cohorts between 3 to 6 patients starting at a dose of 0.025 mg/kg with escalation or de-escalation.
  The aim of this Phase 1b study is to investigate the safety and fluorescence signal of a single dose of LS301-IT, a novel fluorescence imaging agent developed by Integro Theranostics (IT), administered by slow intravenous (IV) in patients undergoing surgical thoracoscopy and VATS (Video-Assisted Thoracoscopic Surgery) resection of lung cancer. Safety is the primary objective of this study, followed by evaluation of the fluorescence signal as it relates to dose level and dosing time interval which will not be used for decision-making in the surgical resection in this study.
Who Masked: Outcomes Assessor
Masking Description: The pathologist evaluating the biopsy samples will be blinded as to patient participation in the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- LS301-IT Cohort -1 (Experimental): 0.0125 mg/kg LS301-IT administered by IV infusion over approximately 15 minutes the day before surgery
  Interventions: Drug: LS301-IT
- LS301-IT Cohort 1 (Experimental): 0.025 mg/kg LS301-IT administered by IV infusion over approximately 15 minutes the day before surgery
  Interventions: Drug: LS301-IT
- LS301-IT Cohort 2 (Experimental): 0.05 mg/kg LS301-IT administered by IV infusion over approximately 15 minutes the day before surgery
  Interventions: Drug: LS301-IT
- LS301-IT Cohort 3 (Experimental): 0.075 mg/kg LS301-IT administered by IV infusion over approximately 15 minutes the day before surgery
  Interventions: Drug: LS301-IT

INTERVENTIONS:
Drug: LS301-IT — LS301 is composed of: 1) a cyclic peptide that binds phosphorylated Annexin A2 (ANXA2) which is found on the surface of malignant cells typically located in solid tumors and in malignant lymph nodes; and 2) cypate, a near infrared (NIR) molecule conjugated to the peptide, which fluoresces when illuminated using NIR light.

SUMMARY:
The aim of this Phase 1b study is to investigate the safety and fluorescence signal of a single dose of LS301-IT, a novel fluorescence imaging agent developed by Integro Theranostics (IT), administered by slow intravenous (IV) administration in patients undergoing surgical thoracoscopy and resection of lung cancer. Safety is the primary objective of this study, followed by the evaluation of the fluorescence signal as it relates to dose level and dosing time interval.

DETAILED DESCRIPTION:
This is a Phase 1b, open-label study to investigate the use of LS301-IT (investigational medicinal product [IMP]), a fluorescence imaging agent used for visualization of tumor margins and other suspicious nodules in patients with primary diagnosis, or a high clinical suspicion, for cancer in the lung based on CT, biopsy, or other imaging.

Up to 24 patients (4 dose cohorts, up to 6 patients each) for Phase 1b study (total of 24 patients maximum). There will be no stratification by dosing interval or lung cancer type (e.g., lung adenocarcinoma, lung squamous cell carcinoma).

As safety is the primary objective of this study, the safety of each dose level will be assessed by the Safety Review Committee (SRC). Based upon the safety results of the first cohort, the SRC will recommend to the Sponsor which dose levels of LS301-IT may be administered in subsequent cohorts.

ELIGIBILITY:
Inclusion Criteria:

* ECOG performance status of 0 to 2
* Have a primary diagnosis, or a high clinical suspicion, for cancer in the lung based on CT, biopsy, or other imaging.
* Are scheduled to undergo surgical thoracoscopy and resection of the lung.

Exclusion Criteria:

* Contraindications for surgery or any medical condition that in the opinion of the investigator could jeopardize the safety of the subject
* No planned surgical use of any other fluorescent optical imaging agent, or exposure to another optical imaging agent within 8 weeks prior to surgery

History of any drug-related hypersensitivity or anaphylactic reactions, including those attributed to indocyanine green (ICG) or other agents used in the study, or known shellfish allergies.

Known sensitivity to near infrared light

Patients with impaired renal function as defined by a creatinine clearance (CrCl) <60 mL/min at Screening, according to the Cockcroft-Gault formula ((140 - age) × body weight/plasma creatinine × 72 (× 0.85 for female)

History, or presence in the ECG at Screening, of any clinically significant abnormalities including cardiac conduction abnormalities such as Fridericia's corrected QTc interval (QTcF) > 470 ms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-11-07 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Number of Patients with Dose Limiting Toxicities | 2 to 7 days after dosing
  Dose Limiting Toxicity - Any CTCAE Grade 2, 3, 4, or 5 AE (any treatment emergent sign or symptom) at least possibly related to IMP will be considered a DLT, as well as any other AE deemed clinically relevant by the SRC.
Number of Patients that discontinue the study or have their surgery cancelled due to toxicity | From start of dosing to time of surgery
  Treatment discontinuation and/or surgery cancellation due to toxicity (hypersensitivity reaction to LS301-IT)

OTHER OUTCOMES:
Maximum observed plasma concentration (Cmax) in ng/mL | Samples collected up to 24 hours after dosing
  Cmax of LS301 and its main metabolite
Area under the plasma concentration time curve from time 0 extrapolated to infinite time (AUC0-∞ [AUCinf]) in ng*hr/mL | Over 24 hours after dosing
  AUC of LS301 in plasma.
Area under the plasma concentration-time curve from time 0 to the last quantifiable plasma concentration (AUC0-t [AUClast]) in ng*hr/mL | over 24 hours after dosing
  LS301 concentration in plasma
Time to reach maximal plasma concentration (Tmax) in minutes | over 24 hours after dosing
  LS301 concentration in plasma
Elimination/apparent terminal elimination half- life (t1/2) in minutes | 24 hours after dosing
  LS301 concentration in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Robert Honigberg, MD, Study Director — Integro Theranostics
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided